## **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

MEDICAL RECORD

Adult Patient or
 Parent, for Minor Patient

INSTITUTE: National Institute of Allergy and Infectious Diseases

STUDY NUMBER: 13-I-0141 PRINCIPAL INVESTIGATOR: Michael C. Sneller, MD

STUDY TITLE: A Phase I Randomized, Double-Blind, Placebo-Controlled Study of a Multi-Antigen DNA Vaccine

Prime Delivered by In Vivo Electroporation, rVSV Booster Vaccine in HIV-Infected Patients Who

Began Antiretroviral Therapy During Acute/Early Infection

Continuing Review Approved by the IRB on 03/09/15

Amendment Approved by the IRB on 08/19/15 (F)

Date Posted to Web: 08/29/15

Standard

## **INTRODUCTION**

We invite you to take part in a research study at the National Institutes of Health (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in at least one study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

## **PURPOSE OF THE STUDY**

You are invited to participate in this study because you:

- Are infected with the human immunodeficiency virus (HIV), and
- Began your HIV treatment shortly after becoming infected, and
- Are currently on an HIV-treatment regimen and are willing to interrupt your HIV treatment for 16 weeks

#### PATIENT IDENTIFICATION

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or • Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

File in Section 4: Protocol Consent (1)

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141 CONTINUATION:  pages

In most people infected with HIV, their immune system (the body's normal ability to fight off disease) can't control or cure the infection. Combination antiretroviral therapy ('cART' – a combination of anti-HIV drugs taken daily) can keep the amount of HIV virus very low for a long time. However, if treatment is stopped, the immune system isn't able to control the infection, and HIV levels go up again. Also, cART doesn't completely remove HIV from your body.

The purpose of this study is to see how well people with HIV tolerate "therapeutic vaccination." Therapeutic vaccination means giving a vaccine to TREAT an infection that someone already has (HIV in this case). Normally, we give vaccines to PREVENT a person from getting infections (for example, there are vaccines to prevent the flu and the measles).

We also want to see how levels of HIV, CD4 cells (the 'good' immune cells that are damaged by HIV), and other measures of HIV infection change after a person receives this vaccination. We plan to show this by stopping cART after some people have been given therapeutic vaccination and others have been given a placebo (a salt water-like solution that should have no effect), for comparison.

Therapeutic vaccination in this study is produced by Profectus BioSciences and includes 2 different investigational vaccines against HIV (HIV-MAG pDNA and VSV HIV *gag*). The HIV-MAG pDNA vaccine will be combined with an investigational 'adjuvant' (a substance that should make vaccines more potent) called IL-12 pDNA. The HIV-MAG pDNA and adjuvant will be given by an investigational device to inject the vaccines into the muscle in your arm. This injection method is called electroporation (EP) and is designed to improve how well your body absorbs some vaccines.

The study vaccines, adjuvant, and EP injection device have not been approved by the Food and Drug Administration (FDA); they will be used in the current study with permission from the FDA for experimental use. That means we don't know whether they are safe to use in people, or whether they will work to treat your HIV infection.

## **STUDY VACCINES**

<u>HIV-MAG pDNA (HIV-MAG)/IL-12 pDNA adjuvant (adjuvant)</u>: The HIV-MAG vaccine contains some DNA (genetic material required for cells to function) made in the laboratory. The particular DNA in the study vaccine tells the body to make proteins that are normally found in HIV. It is hoped that making these non-infectious proteins will trigger your body to better fight the 'real' HIV that you have.

The HIV-MAG vaccine is being given with an adjuvant also made of DNA, which we hope will stimulate your body to make IL-12 proteins, which also help fight infection.

**VSV HIV** gag (VSV): This vaccine will be given to you at 2 time points during the trial, after the HIV-MAG, to try to further strengthen your immune response against HIV. VSV carries some DNA that tells your body to make another protein that is found in HIV, which may give your body another 'target' to attack on 'real' HIV in your system.

The VSV vaccine is made from a virus normally spread to animals by insect bites. Infected animals may get a rash or sores at the location of the bite, around the mouth, or on their hooves, which go away within 10-12 days. Human infection with natural VSV is very rare and can produce a mild self-limited disease similar to that seen in animals.

**PATIENT IDENTIFICATION** 

**CONTINUATION SHEET for either:** 

NIH-2514-1 (10-84) NIH-2514-2 (10-84) P.A.: 09-25-0099

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141 CONTINUATION:  pages

The VSV in the current study vaccine has been weakened so that it can't cause the health problems seen in animals. It is very unlikely that someone who receives the study vaccine will develop any symptoms of VSV infection or pass VSV to someone else.

## WHO WILL BE IN THE STUDY

A total of 30 people, 18 to 65 years of age, with HIV are expected to be enrolled in this study. To be in the study, you must be willing to stop your HIV treatment for about 16 weeks during the study period and, if you are sexually active, you and your partner must agree to take steps to help reduce the chance of passing on the HIV infection, or of pregnancy.

#### STUDY SCHEDULE

Your study participation time is expected to be about 26 months. Some visits need to be at the NIH Clinical Center in Bethesda, Maryland, and some may possibly be done closer to your home. The study staff will let you know what to expect in your case.

Screening visit: About 1 to 2 months before the first (baseline) study visit, you will be asked to sign this informed consent document, and then you will have the following procedures done over 1 or 2 days:

- Physical exam, medical history, medication list, electrocardiogram (EKG or ECG).
- Test for body fat content, done by a 'skin-pinch' test.
- Blood and urine collection, including a pregnancy test and other testing related to HIV and your general health.

During the screening visit and throughout the study until the visit at week 56, you will continue to take HIV medications (cART).

Baseline visit: If you are eligible to participate, you will return for a baseline study visit. You will be randomly assigned (by chance, like flipping a coin) to receive EITHER the vaccines we are trying to study (HIV-MAG, adjuvant, and VSV) or a placebo ('pretend' vaccine that is made of salt water, so it should not have any medical effect). Neither the study staff nor you will know your group assignment until after the study is completed.

The visit will occur over 1 to 3 days for about 2 to 5 hours each day. Before receiving the vaccination, you will have medical procedures that are similar to those done at the screening visit (above) as well as:

- Leukapheresis (collection of your white blood cells for the study).
- Instructions on the use of a diary card.

After the study procedures, you will receive the first dose of the study vaccine (HIV-MAG and adjuvant) or the placebo vaccine; these will be delivered with the EP device, which is described in the risk section of this document. The study doctor will then evaluate you for symptoms related to the vaccine.

P.A.: 09-25-0099

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141 CONTINUATION:  pages

**Vaccination-phase visits:** During week 4 through week 56, you will come in for 10 study visits. Each visit will take about 2 to 3 hours to complete, except for the visits at week 36 and 56, which will take about 2 to 5 hours to complete. Depending on your group assignment, you will be administered again either the HIV-MAG pDNA vaccine and IL-12 pDNA adjuvant or the placebo vaccine during the visits at week 4, 12, and 36. In addition, you will receive the other study vaccine (VSV HIV *gag*) or the placebo vaccine during the visits at week 24 and 48.

During the visits at week 4, 12, 24, 36, 48, and 56, you will have the routine medical procedures and other procedures done, including:

- Physical exam, medical history, medication list.
- Vital signs.
- Blood draw.
- Blood or urine pregnancy test.
- Leukapheresis (at week 36 and 56 only).
- Evaluation of vaccine-related symptoms (at week 4, 12, 24, 36, and 48 only).
- Evaluation of any new symptoms.
- Evaluation of your diary card.
- Oral swabs—only in individuals who develop mouth sores.

In addition, you will have your blood drawn again during the visits at week 14, 26, 38, and 50.

<u>Treatment-interruption phase visits</u>: During week 58 through week 72, you will come in every 2 weeks for 7 study visits; each visit will take about 1 hour to complete.

After the study visit at week 56, you will stop your HIV treatment until the visit at week 72. If you are taking any non-nucleoside reverse transcriptase inhibitors (NNRTIs; for example, Rescriptor, Sustiva, or Viramune), the NNRTI will be switched to another HIV drug that is either a protease inhibitor (for example, Reyataz or Prezista) or an integrase inhibitor (for example, Isentress) for about 2 weeks before stopping your HIV treatment. This is to prevent the development of resistance to the NNRTI drugs that can potentially occur because these drugs tend to stay in your body longer than the other HIV drugs.

Your blood will be drawn every 2 weeks during each study visit. If you live outside the local Bethesda, Maryland area, you may be asked to go to your local physician for the blood draws; the study doctor will discuss this possibility with you.

During the visits at week 64 and 72, in addition to the blood draw, you will also have the following procedures done:

- Physical exam with review of medical history.
- Vital signs.
- Evaluation of any new symptoms.

If you develop HIV-related symptoms, your viral levels go up to high levels for more than 4 weeks, or your CD4 cell counts (a type of white blood cells) decrease to low levels, you will return to the NIH Clinical Center for an additional visit to be evaluated. If the study doctor determines that you can't continue without your HIV treatment, you will be restarted

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141

CONTINUATION:  pages

on your HIV treatment and will be followed for 6 months. Also, you will undergo the procedures listed under the study visits at week 84 and 96 below.

If you and your private physician decide to restart your HIV treatment, you can choose any combination of drugs for the HIV treatment. You should call the study team for an appointment **BEFORE** you restart any HIV treatment. We would like to collect additional blood from you before you restart the HIV treatment.

**Follow-up phase:** During week 76 through week 96, you will come in every month for 4 study visits; each visit will take about 1 to 2 hours to complete.

After the visit at week 72, you will restart your HIV treatment and will continue on it through week 96 (end of study). Following the week 96 visit you will have completed the study and return to the care of your home physicians.

During the follow-up phase, your blood will be drawn every month until the level of HIV in your blood is suppressed. If you live outside the local Bethesda, Maryland area, you may be asked to go to your local physician for the blood draws; the study doctor will discuss this possibility with you.

During the visits at week 84 and 96, in addition to the blood draw, you will also have the following procedures done:

- Physical exam with review of medical history.
- Vital signs.
- Evaluation of any new symptoms.

#### STUDY PROCEDURES

**Physical exam with medical and medication history:** You will be evaluated by the study staff and will undergo a physical exam. You will be asked about how you are feeling, if you've had any illness recently, and about the medications you are taking now and have taken in the past, including non-prescription drugs. A weight measurement will also be done at some of the visits.

<u>Vital signs</u>: Your blood pressure, heart rate, respiratory rate, and temperature will be recorded.

**Skin-pinch test:** This test will be done to measure the thickness of the skin on your upper arm muscles for the administration of the study vaccines.

Vaccine injection with the EP device: The HIV-MAG pDNA/IL-12 pDNA adjuvant and the placebo vaccine will be injected with an investigational EP device, which is a small, hand-held tool. The device will be pressed against your upper arm firmly, and the injection needle will then be inserted into your arm, and the contents of the study vaccine/ placebo vaccine will be delivered through the needle 3 to 4 seconds later. After the injection, a very small amount of electricity will be sent through your arm muscle. You may feel some mild pain or discomfort, which goes away quickly for most people. This procedure will be done once in each upper arm for each of the HIV-MAG pDNA/IL-12 pDNA vaccinations.

**Blood draw:** Blood will be drawn from a vein in your arm to measure your blood cell counts, to see if your organs are working well, including your liver and kidneys, and to measure your HIV levels; your blood will also be used to test for

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141 CONTINUATION:  pages

hepatitis B and C, which cause liver disease, and for syphilis, which is a sexually transmitted disease. The total volume of blood collected during the study will not exceed the guidelines for blood collected for research in adult subjects at the NIH Clinical Center. While in the study, let the study team know if you are participating in other studies or have blood drawn for any other reason.

**<u>Urine collection</u>**: A sample will be collected for routine laboratory tests.

**Blood or urine pregnancy test:** For women of childbearing potential, a pregnancy test will be done using a blood or urine sample. You will not be allowed to participate in the study if you are pregnant.

**EKG**: This test records the normal electrical activity of your heart. Electrodes, which are soft, sticky patches attached to wires, will be placed on the skin of your chest, arms, and legs. The procedure does not cause any pain or harm.

**Leukapheresis:** For this procedure, some blood will be removed through a needle in your arm, your white blood cells will be separated from the blood, and the rest of the blood will be returned to your body through another needle. Citrate, a generally harmless chemical to prevent blood from clotting in the machine, will still be in the blood that returns to you. This procedure will be done in the Department of Transfusion Medicine at the NIH Clinical Center. You will be asked to sign a separate consent form that will describe in more detail how the procedure will be done and the risks associated with it.

Leukapheresis provides us with many more white blood cells than we could get from a routine blood draw, but this will still be a small fraction of the total number in your body. The body quickly replaces the cells that were removed. The procedure will take approximately 1 to 3 hours to complete. A doctor will be available in or near the leukapheresis clinic at all times.

**Evaluation of vaccine-related symptoms/diary cards:** After each vaccination, you will have to wait at the clinic for about an hour to see if you experience any symptoms related to the vaccine. You will be asked to write down how you feel and your symptoms in a diary card, which will be given to you during the baseline visit. After you receive the study vaccine at week 0, 4, 12, and 36, you will be asked to record your symptoms during the first night and the following 3 days; after you receive the VSV study vaccine at week 24 and 48, you will be asked to record your symptoms during the first night and the following 7 days. During these times, you will also be asked to contact the study team at the NIH Clinical Center daily.

The diary card will take you about 10 minutes to complete each day. You will be asked to bring the diary card back to the clinic during your next visit, and it will be collected by the study staff. If you stop the study early, the diary card will be collected during your last visit.

You must contact the study staff if you have any issues or concerns after receiving the vaccinations. If you have a problem, we will continue to evaluate you until it goes away.

<u>Oral swabs</u>: Individuals who develop mouth sores up to 7 days after injection with the VSV HIV *gag* vaccine will have samples collected from their sores to test for VSV infection.

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141

CONTINUATION:  pages

## RISKS ASSOCIATED WITH THE STUDY

<u>General risks associated with vaccines</u>: Possible risks associated with vaccines include fever, chills, rash, aches and pains, nausea, headache, dizziness, and fatigue. We know these side effects can occur with other vaccines. They can occur if you receive the study vaccines or the placebo vaccine in this study. The side effects don't usually last long.

As with all vaccines or drugs, you could have an immediate allergic reaction, including itchy rash, hives, low blood pressure, sudden body swelling, or even difficulty breathing. Allergic reactions can be life threatening; therefore, the study staff will watch you for 1 hour after each vaccination. There may be other side effects, even serious ones that we don't yet know about. Therefore, it is important that you report all the side effects to the study staff as soon as they occur.

Very rarely, vaccines may cause your immune system to attack your own body and blood cells. We don't know the risk for having this kind of "auto-immune" problem due to the study vaccines.

Risks associated with the HIV-MAG pDNA vaccine/IL-12 pDNA adjuvant: We don't know all the risks associated with the HIV-MAG pDNA study vaccine because it has only been given to about 150 people. Possible risks related to similar DNA vaccines include muscle damage at the site of the injection, "auto-immune" problems (see the paragraph, above), or vaccine DNA mixing with your own DNA. This could lead to cancer or unknown side effects. We think the risk of these things happening is very low. In other studies, more than 1,000 people have been given DNA vaccines being tested against HIV and none of these things has happened so far. We expect the risks of the HIV-MAG pDNA vaccine in this study to be similar to those of other HIV DNA vaccines. However, there may be new side effects that we don't yet know about.

In earlier studies of the IL-12 pDNA adjuvant, there have been no severe side effects related to the adjuvant. We don't know if participants in this study will have similar side effects to those seen in earlier studies.

**Risks associated with bupivacaine:** The HIV-MAG pDNA vaccine and IL-12 adjuvant contain bupivacaine. It is a numbing medicine similar to that used by dentists. At much higher doses, bupivacaine and other medications in the same group of local anesthetics can cause serious problems with the nervous system (brain, spinal cord, nerve cells) and the heart. Other possible side effects include nausea, vomiting, chills, rash, hives, difficulty breathing, and severe allergic reactions. However, in this study, we will be using doses about 10 times lower than the dose that has been known to cause these side effects.

**Risks associated with the EP device:** An injection with the EP device will cause brief muscle contractions during the procedure. In previous studies using EP, people often felt an initial pain that ranged from mild to moderate. For most people, the pain eased quickly (within an hour). EP can also cause soreness, bruising, redness, swelling, itching, or hardness/stiffness in the upper arm where you got the injection. A standard vaccine injection (such as tetanus or flu vaccine) with an ordinary needle and syringe can also have these same side effects.

Other unlikely but possible side effects include:

- Infection at the injection site.
- Abnormal heart rhythm.

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141 CONTINUATION:  pages

• Damage or malfunction of pacemakers, and other metal medical materials in the body. You cannot be in the study if you have heart problems, or have metal medical devices in the upper body or arms.

The EP device has been used in about 280 people so far, and no serious side effects have been observed.

Also, we don't know if the EP device will increase the risks associated with any of the study products.

Risks associated with the VSV HIV gag vaccine: VSV in the study vaccine has been weakened so that it doesn't cause the illness seen in animals. However, it is still possible, although very unlikely, that the study vaccine could cause symptoms that people get from VSV infection, including fever, muscle aches, headaches, fatigue, encephalitis, or mouth sores. Encephalitis is a brain disease that can cause confusion, drowsiness, seizures, and loss of consciousness. Only 1 person (a young child) is reported to have developed possible encephalitis that was possibly caused by natural VSV infection. The weakened virus used to make the VSV vaccine for the current study is not expected to cause encephalitis. In trials of healthy adults, immunization with the VSV vaccine has been found to be associated with self-limited sores in the mouth and a transient (less than 2 days) decreases in lymphocyte counts in some individuals. If you notice sores in your mouth, please notify the study team immediately so they can arrange for a mouth swab to look for the VSV virus.

Because the VSV vaccine has only been given to about 60 people so far, there might be other risks associated with this vaccine that we don't yet know about.

Risks associated with treatment interruption: People who started HIV treatment early in their infection may have stronger immune responses to the virus. These immune responses cannot control the infection in the vast majority of people and treatment with anti-HIV drugs is needed. The long-term effects, if any, of temporarily stopping your HIV treatment are not yet known. It is possible that your CD4 cell counts may decrease, your HIV disease may get worse, or the number of cells in which the virus remains latent (hidden or resting) may increase. Studies of temporarily (for 4-6 months) stopping HIV treatment in individuals treated during early infection have not found decreases in immune function or long-term problems. However, there might be risks of temporarily stopping your HIV medications that we don't yet know about. We will monitor your CD4 cell counts and viral levels closely during the 16-week period when you will be off treatment.

Another possible risk associated with stopping your treatment includes drug resistance. "Drug resistance" means that a drug given to treat HIV no longer works against it. This is a special concern if you are currently taking NNRTIs because these drugs tend to remain in the body longer than other drugs do, which could increase the risk of making the virus resistant to that drug or other NNRTI drugs. If you are taking any NNRTI drugs, you will be switched to a protease inhibitor or an integrase inhibitor about 2 weeks before stopping your HIV treatment to minimize this risk.

There may be an increased risk of transmitting HIV (for example, to a sexual partner who does not have HIV) during the treatment interruption if your viral levels increase during this time. However, it is important to realize that even while taking HIV treatment you can still pass the HIV virus to others by sexual contact. So, "safe-sex practices" should always be used. A member of the study team will review safe-sex practices with you prior to study enrollment and again prior to the treatment interruption.

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141 CONTINUATION:  pages

**Risks associated with the study vaccines during pregnancy:** It is not known how the study vaccines will affect a developing baby. Therefore, if you are a woman of childbearing potential, you must agree to use 2 acceptable methods of contraception (birth control pills, male/female condoms, diaphragm or cervical cap, or intrauterine device) beginning at least 3 weeks before the first dose of the study vaccine/placebo vaccine and continuing until your last study visit.

**Risks associated with leukapheresis:** Donations for this procedure are generally safe and side effects are rare. Pain, bruising, or discomfort at the needle injection site may occur. Sometimes leukapheresis can cause a tingling sensation around the mouth or in the finger, chills, nausea, heartburn, or mild muscle cramps. These side effects can usually be relieved by slowing or temporarily stopping the leukapheresis or taking a calcium-containing antacid, such as Tums. Other possible side effects are anxiety, vomiting, and lightheadedness. Temporary lowering of your blood pressure may also develop. On rare occasions, fainting or seizure may occur. Very rarely, a nerve problem at the needle injection site may occur, or malfunction of the machine used for the procedure may occur, resulting in a loss of about one pint of your blood.

There are possible risks from re-infusion of the blood after being processed by the machine, such as infection or a side effect from the blood components. However, this has not been seen in many thousands of volunteers who have undergone this or similar procedures to date.

**Risks associated with HLA testing:** Some of the blood drawn from you as part of this study will be used for a test for HLA type, which is a genetic test for markers of the immune system. It is usually used to match bone marrow or organ transplants. For research, HLA testing might be used to try to identify factors associated with the progression of disease or related conditions. In addition, determining the HLA type is necessary to perform certain research studies. Results from the HLA testing will become a part of your medical record at the NIH. Medical records containing this information are maintained in a secured manner. Although we are committed to confidentiality, a court could still subpoena your medical records. All of these issues should be carefully considered before joining the study.

<u>Risks associated with the blood draw</u>: The risks associated with drawing blood from a vein in your arm include pain, bruising, and, rarely, infection at the site, hematoma or black and blue mark with a lump caused by blood release into the tissues, lightheadedness, and fainting.

## **BENEFITS ASSOCIATED WITH THE STUDY**

It is possible that you may get a treatment that will improve your immune response against your HIV infection, which may help to control it better. It is also possible that you may receive no benefit from participating in this study. Information learned from the study may help others infected with HIV.

## **ALTERNATIVES TO PARTICIPATING IN THIS STUDY**

You may choose not to participate in this study and continue to receive care from your current physician(s) or enroll in other clinical studies.

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141

CONTINUATION:  pages

#### WITHDRAWAL FROM THE STUDY

You can stop participating in this study at any time. Tell a member of the study team if you no longer want to participate. Samples and data collected prior to this request will be stored for the duration of the protocol unless you specifically request the removal of all your samples from the study.

If you decide to leave, we may ask you to return for a final visit to perform some tests and exams to ensure safety. However, you will not be required to return for this visit. If you stop taking the study vaccine before the visit at week 24, you will continue to be followed for safety purposes; but, you will not be required to stop your HIV treatment after the visit at week 56.

If you choose to withdraw your participation in the study, this will not affect your participation in other clinical trials at the NIH.

## **EARLY REMOVAL FROM THE STUDY**

You may be removed from this study early without your consent for the following reasons:

- You enroll in another clinical study of an experimental treatment.
- You develop a health problem, an abnormal lab test, or any medical disease that, in the opinion of the study doctor, puts you at increased risk of harm or it's not in your best interest.
- You become pregnant.
- You miss more than 1 vaccination.
- You repeatedly miss the study visits or refuse to comply with the study guidelines or procedures.
- You exhibit inappropriate or threatening behavior towards NIH staff or other subjects.
- If the study is stopped or cancelled.

•

#### **COMPENSATION**

You will receive financial compensation for the leukapheresis procedure according to the NIH Clinical Center volunteer guidelines: \$100.00 for a 2-pass leukapheresis procedure or \$200.00 for a 4-pass leukapheresis procedure. The study doctor will let you know which procedure you're having done.

## **COSTS ASSOCIATED WITH THE STUDY**

There will be no charge to you or your health insurance company for any of the tests, procedures, or medications that are directly related to this study. The costs for any other medical care provided outside the NIH during this period will not be covered.

#### **NEW FINDINGS**

Any new findings discovered during this study that are considered relevant to your health or to your decision to continue in the study will be fully discussed with you.

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 13-I-0141

CONTINUATION:  pages

## STORED SAMPLES/DATA AND FUTURE RESEARCH

If you agree to participate in this study, you also agree to let us store your blood samples and data for future research. The stored samples/data may help us learn more about the effect of the HIV-MAG pDNA/IL-12 pDNA adjuvant and the VSV HIV *gag* vaccine on HIV infection. The samples/data will be labeled with a code that only the study team can link to you. Any information that can be traced back to you will be kept as private as possible. If you change your mind and decide you do not want us to store your samples, please contact us. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy all your samples.

Your coded samples/data might be sent to other study doctors for their research. Other information, such as your sex, age, health history, or ethnicity might also be shared. Your samples will not be sold, and you will not be paid for any products that result from this research. Future studies may require health information about you, such as smoking history or present health status, which we don't already have. If so, our study team may contact you. Future research that uses your samples/data will not help you, but it may help us learn more about HIV infection and other health problems. In general, the research tests performed in this study are not like routine medical tests, and they may not relate directly to your medical care.

#### **CONFLICT OF INTEREST**

The NIH reviews its staff researchers at least yearly for conflicts of interest. You may ask your study team for additional information or a copy of the Protocol Review Guide. This protocol has investigators who are not NIH employees. Non-NIH investigators are expected to adhere to the principles detailed in the Protocol Review Guide, but they are not required to report their personal financial holdings to the NIH. Profectus Biosciences is providing the vaccines for this study to NIH without charge. No NIH employee involved in this study receives any payment or other benefits from Profectus Biosciences.

## **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

• Adult Patient or • Parent, for Minor Patient

STUDY NUMBER: 13-I-0141 CONTINUATION:  pages

## OTHER PERTINENT INFORMATION

1. Confidentiality. When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- **2. Policy Regarding Research-Related Injuries.** The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- **3. Payments.** The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH guidelines.
- **4. Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Dr. Michael Sneller, Building 10, Room 9N208, Telephone (301) 496-0491. You may also call the Clinical Center Patient Representative at (301) 496-2626.

**5. Consent Document.** Please keep a copy of this document in case you want to read it again.

| COMPLETE APPROPRIATE ITEM(S) BELOW: | |
|---|---|
| A. Adult Patient's Consent | B. Parent's Permission for Minor Patient. |
| I have read the explanation about this study and have been | |
| given the opportunity to discuss it and to ask questions. I | |
| hereby consent to take part in this study. | hereby give permission for my child to take part in this study. |
| | (Attach NIH 2514-2, Minor's Assent, if applicable.) |
| | (Attach Min 231 i 2, Minor 3 Assent, ii applicable.) |
| Signature of Adult Patient/Legal Representative Date | Signature of Parent(s)/Guardian Date |
| Print Name | Print Name |
| C. Child's Verbal Assent (If Applicable) | |
| The information in the above consent was described to my child and my child agrees to participate in the study. | |
| Signature of Parent(s)/Guardian Date | Print Name |
| Dute Dute | Time Name |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE | |
| FROM MARCH 9, 2015 THROUGH MARCH 8, 2016. | |
| Signature of Investigator Date | Signature of Witness Date |
| Signature of investigator Date | Signature of whitess |
| Print Name | Print Name |

## **PATIENT IDENTIFICATION**

# **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)**

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent